CLINICAL TRIAL: NCT00005544
Title: Community Based Study of Adult Onset Asthma
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5087; R01HL061302 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-05

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To identify the role of irritant exposure in adult-onset asthma by simultaneously using both clinical and case control methods in a community-based perspective study of asthma incidence.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma incidence is increasing, and in adults work-related exposures may be an important factor-occupational asthma (OA) incidence increased 70 percent over the last decade according to a recent registry based study. The true contribution of occupational exposures to adult-onset asthma is unknown because the methods for measuring OA give conflicting results. Methods based on surveillance of clinically diagnosed OA account for less than one to five percent of adult-onset asthma. However, case-control methods of measuring asthma risk by industry suggest that six to 33 percent of adult-onset asthma is caused by workplace exposures. The conflict may occur because of two factors: physicians often fail to diagnose and report OA, and irritant exposures may increase the risk the risk of asthma without causing cases that meet the clinical definition. Both factors have important implications for proper treatment and prevention of asthma in adults.

DESIGN NARRATIVE:

Clinical and case control methods were used to identify the role of irritant exposure in adult-onset asthma in a community-based prospective study of asthma incidence. The study cohort was a typical US working population enrolled in an HMO. Additional benefits of the study design were the opportunities to validate a questionnaire for exposure assessment and for detection of work-related asthma. Specifically, the study: 1) Investigated incident cases in a cohort of over 80,000 adults over three years and determined the proportion that met a clinical definition of occupational asthma (OA); 2) Used a nested case-control study to determine the incidence of all asthma by occupation and workplace exposure; 3) Determined whether clinical OA accounted for the excess incidence of adult-onset asthma associated with workplace exposure to sensitizers and irritants; 4) Prospectively followed asthmatics for two years after diagnosis to determine the impact of adult-onset asthma on lung function, employment, income, and quality of life, and to determine whether prognosis differed for clinical OA and for asthma associated with workplace irritant exposure; 5) Tested an intervention designed to increase appropriate clinical diagnosis, and thus secondary prevention of OA.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-02; Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Milton — Harvard University School of Public Health

REFERENCES:
- [Background] Sama SR, Hunt PR, Cirillo CI, Marx A, Rosiello RA, Henneberger PK, Milton DK. A longitudinal study of adult-onset asthma incidence among HMO members. Environ Health. 2003 Aug 7;2(1):10. doi: 10.1186/1476-069X-2-10. PMID 12952547